CLINICAL TRIAL: NCT00768040
Title: A Randomized, Double-masked, Placebo-controlled, add-on Study to Assess the Efficacy of Oral Aliskiren 300 mg Once Daily for Diabetic Macular Edema
Brief Title: Efficacy of Aliskiren in the Treatment of Diabetic Macular Edema
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPP100A2244; EudraCT 2008-00581-23
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-02

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes; Macular edema; Aliskiren; Diabetic retinopathy; Diabetes mellitus type 1; Diabetes mellitus type 2
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema; Diabetic Retinopathy; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren 300 mg (Experimental): Aliskiren 300 mg once daily for 12 weeks
  Interventions: Drug: Aliskiren
- Placebo (Placebo Comparator): Matching placebo once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — 300 mg once daily
  Other Names: SPP100
  Arms: Aliskiren 300 mg
Drug: Placebo — Matching placebo once daily
  Arms: Placebo

SUMMARY:
To assess the efficacy of oral aliskiren as a therapy for diabetic macular edema

ELIGIBILITY:
Inclusion criteria:

* Type 1 or type 2 diabetes
* Diabetic macular edema

Exclusion criteria:

* Recent intra-ocular surgery in the study eye (e.g., cataract surgery in the last 6 months)
* Recent laser photocoagulation in the study eye
* Recent treatment with Avastin, Lucentis, or intravitreal corticosteroids in the study eye

Other protocol-defined inclusion/exclusion criteria applied

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (10):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina-Vitreous Associates, Los Angeles, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Georgia Retina, Atlanta, Georgia
  - Elman Retina Group, Baltimore, Maryland
  - Joslin Clinic, Boston, Massachusetts
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Charlotte Eye, Ear, Nose and Throat Associate, Charlotte, North Carolina
  - Retina-Associates of Cleveland, Inc, Beachwood, Ohio
  - Retinal Consultants of Houston, Houston, Texas
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren 300 mg | Placebo
Started | 20 ("Started" indicates randomized, safety and full analysis set.) | 19
Completed | 16 | 16
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 2
Not completed — Abnormal laboratory value | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 300 mg | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.76) | 60.1 (10.57) | 62.2 (10.74)
Age, Customized [Number; unit: participants]
  18 - 64 years | 9 | 13 | 22
  65 - 84 years | 11 | 6 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Retinal Thickness in Patients With Type 1 or Type 2 Diabetes, After 12 Weeks of Treatment
Description: The central retinal thickness was measured by Optical coherence tomography (OCT). The changes in central retinal thickness (CRT) from baseline to the end of study at week 12 were analyzed using a univariate analysis of covariance model (ANCOVA) with baseline value as a covariate and treatment as a fixed factor
Time Frame: Baseline to week 12
Population: This study was terminated early due to low recruitment of patients.
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Aliskiren 300 mg | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Aliskiren 300mg: Aliskiren 300 mg once daily for 12 weeks
Arm/Group | Aliskiren 300mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/19
Other Adverse Events (participants affected / at risk) | 13/20 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300mg (N=20) | Placebo (N=19)
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300mg (N=20) | Placebo (N=19)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Cataract subcapsular (Eye disorders) | 0 | 1
Choroidal neovascularisation (Eye disorders) | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0
Hyalosis asteroid (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 1 | 1
Retinal exudates (Eye disorders) | 0 | 1
Retinal neovascularisation (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early due to low recruitment of patients. The study lacked power against the original objective of statistically significance for changes in central retinal thickness due to the much reduced sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.